



## Measurement and Validation of Fetal Heart and Fetal Movement Signals Detected via Non-adhesive Sensors – Second Phase

## **Consent Form**

If you are happy to participate please complete and sign the consent form below

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet (Version 1.2, Date 03.03.2025) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that my participation in the study is voluntary and that I am free to withdraw at any time without giving a reason and without detriment to myself. I understand that it will not be possible to remove my data from the project once it has been anonymised and forms part of the data set. I agree to take part on this basis. | |
| 3 | I agree to having an ultrasound scan and to monitor my baby's heartbeat with the MONICA AN24 system. | |
| 4 | I understand that my medical records will be accessed by the research team to obtain information relevant to my current pregnancy. | |
| 5 | I agree to having my monitoring session formally observed. | |
| 6 | I agree to having a semi-structured one-to-one interview following the monitoring session. | |
| 7 | I agree to complete a short questionnaire describing my experiences of wearing the sensors and for written responses to be quoted in research reports | |
| 8 | I understand that data collected during the study may be looked at by individuals from The University of Manchester or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my data. | |
| 9 | I agree that any anonymised data collected may be shared with researchers at other institutions. | |
| 10 | I agree that any data collected may be published in anonymous form in academic reports, research websites or journals. | |
| 11 | I agree to take part in this study. | |

## **Data Protection**

The personal information we collect and use to conduct this research will be processed in accordance with data protection law as explained in the Participant Information Sheet and the <u>Privacy Notice for Research Participants</u>.

| Name of Participant | Signature | <br>Date |
|---|---|---|
| Name of the person taking consent | Signature | Date |
| [1 copy for the participant, 1 copy for | the research team (origina | l), 1 copy for the medical notes] |